CLINICAL TRIAL: NCT04559217
Title: Pilot Study of 68Ga-DOTATATE PET/CT and 123I-MIBG Scintigraphy Imaging of Neuroblastoma
Brief Title: 68Ga-DOTATATE Neuroblastoma Imaging Pilot
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-3828
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Neuroblastoma
Keywords: imaging; 68Ga-Dotatate; 68Ga-Octreotate; positron emission tomography (PET)
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Intervention Model Description: Prospective pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm with 68Ga-DOTATATE (Experimental): all participants will undergo a PET scan with 68Ga-DOTATATE
  Interventions: Biological: Radiopharmaceutical 68Ga-DOTATATE

INTERVENTIONS:
Biological: Radiopharmaceutical 68Ga-DOTATATE — Injection of 68Ga-DOTATATE followed by PET/CT acquisition

SUMMARY:
Neuroblastoma is the most frequent extracranial childhood tumor, with an annual incidence of approximately 10.2 per million children. Staging of the disease can be done by different imaging strategies (CT, MRI, scintigraphy and PET/CT). Discrepancies may be observed among these different strategies resulting in different treatment strategies. The goal of this study is to assess the feasibility and safety of 68Ga-DOTATATE and to compare it to 123I-MIBG when investigating neuroblastoma.

DETAILED DESCRIPTION:
Background: Neuroblastoma is the most frequent extracranial childhood tumor, with an annual incidence of approximately 10.2 per million children. Initial staging of the disease and monitoring of the treatment response can be performed with different imaging modalities that include contrast-enhanced computed tomography (ceCT), ultrasound, magnetic resonance imaging (MRI), bone scintigraphy and 123I-MIBG scintigraphy.

Another potential target for neuroblastoma imaging is the somatostatin receptor (SSTR) that is present in many neuroendocrine tumours (NET). The superior PET imaging technology used with new radiotracers (such as 68Ga-DOTATATE) enables imaging at advantageous resolutions well below what is possible by current clinical SPECT systems that are used for 123I-MIBG.

Design: Prospective single-arm non-randomized clinical trial (phase II) - pilot

Objective: 1) Assess the feasibility and safety of 68Ga-DOTATATE PET/CT imaging in patients with neuroblastoma or suspected of having neuroblastoma. 2) Compare lesion-by-lesion the uptake of 68Ga-DOTATATE and 123I-MIBG in the same participant.

Study population: Children and adults with biopsy-proven or suspected neuroblastoma

Procedure and Follow-up: Few days after 123I-MIBG scan, participants will undergo a 68Ga-DOTA-cTATE PET/CT scan (duration 2 hours). Clinical data will be collected from this imaging and from the participant's medical record (demographic, treatment, medication, pathology, lab test results) for a 2-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Newly suspected or biopsy-proven neuroblastoma or recurrence of neuroblastoma
* Planned 123I-MIBG imaging
* Able and willing to provide signed informed consent in French or English (for the adult candidates or the parent/legal tutor of the pediatric candidates)
* Aged between 1 day and 21 years old (inclusively).

Exclusion Criteria:

* History of another cancer in the past 5 years other than non-melanomatous skin cancer.
* Currently under a randomized control trial with unknown allocation;
* Currently under treatment;
* Medical/surgical intervention on the tumour between 123I-MIBG and 68Ga-DOTATATE PET/CT scan.
* Medically unstable or unable to undergo scan.
* Pregnancy (breastfeeding is not an exclusion criterion but needs to be stopped for at least 12 hours after 68Ga-DOTATATE injection).
* Prior allergic reaction to somatostatin analogues

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Accrual rate | For the duration of the study, lasting 6 years
  Number of participants enrolled / year
Rate of adverse events | Up to 24 hours following injection of 68Ga-DOTATATE
  Number of adverse events (being serious or not) associated to the intervention (injection of 68Ga-DOTATATE and PET/CT acquisition

SECONDARY OUTCOMES:
Positive lesions for 68Ga-DOTATATE | One hour post-injection of 68Ga-DOTATATE
  SUV mean of the lesion
Discordance of positive lesions for 68Ga-DOTATATE and positive lesions of 123I-MIBG | Within one week (period between 123I-MIBG scan and 68Ga-DOTATATE scan)
  the number of discordant lesions divided by the number of total positive lesions is the discordance rate

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Rousseau, MD, FRCPC, Principal Investigator — CIUSSSE-CHUS
Locations (3):
- Canada (3):
  - McGill University Health Center - Children's hospital, Montreal, Quebec
  - CHU Ste-Justine, Montreal, Quebec
  - CIUSSS de l'Estrie-CHUS Hospital, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No